CLINICAL TRIAL: NCT01354223
Title: Evaluation of the CooperVision Stenfilcon A Soft Contact Lens for Daily Wear When Compared to the CooperVision Ocufilcon B Soft Contact Lens
Brief Title: Clinical Evaluation of Stenfilcon A Soft Contact Lens When Compared to Ocufilcon B Soft Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FC100239
Record Dates: First submitted 2011-01-10; First posted 2011-05-16 (Estimated); Results first posted 2014-03-21 (Estimated); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Myopia
Keywords: silicone hydrogel contact lens; SHCL; stenfilcon A; ocufilcon B; daily disposable; substantial equivalence; CooperVision ClearSight™ 1 Day SCL
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- stenfilcon A contact lens (Experimental): Randomized to stenfilcon A contact lens worn in a daily wear, daily disposable mode
  Interventions: Device: stenfilcon A contact lens
- ocufilcon B contact lens (Active Comparator): Randomized to ocufilcon B contact lens worn in a daily wear, daily disposable mode
  Interventions: Device: ocufilcon B contact lens

INTERVENTIONS:
Device: stenfilcon A contact lens — Randomized to stenfilcon A contact lens worn in a daily wear, daily disposable mode
  Arms: stenfilcon A contact lens
Device: ocufilcon B contact lens — Daily disposable contact lens worn in a daily wear, daily disposable mode
  Other Names: CooperVision ClearSight™ 1 Day
  Arms: ocufilcon B contact lens

SUMMARY:
This study seeks to evaluate a new daily disposable contact lens compared to an existing daily disposable contact lens.

DETAILED DESCRIPTION:
This study is designed to evaluate the stenfilcon A contact lens to demonstrate substantial equivalence to the Ocufilcon B for market release.

ELIGIBILITY:
Inclusion Criteria:

Prior to being considered eligible to participate in this study, each subject MUST:

* Be at least 18 years of age as of the date of evaluation for the study.
* Have:

  * Read the Informed Consent
  * been given an explanation of the Informed Consent
  * indicated understanding of the Informed Consent
  * signed the Informed Consent document.
* Be willing and able to adhere to the instructions set forth in this protocol and able to keep all specified appointments.
* Be an adapted, current full-time silicone hydrogel or soft contact lens wearer. An adapted full-time wearer is defined as wearing contact lenses on a daily basis for at least 8 hours per day for at least one month prior to participation in the study.
* Possess wearable and visually functional eyeglasses.
* Be in good general health, based on his/her knowledge.
* Require spectacle lens powers between -1.00 and -6.00 diopters sphere with no more than 1.00 diopter of refractive astigmatism and be willing to wear contact lenses in both eyes.
* Have manifest refraction Snellen visual acuities (VA) equal to or better than 20/25 in each eye.
* Upon completing the fitting process with the lenses to be worn in the study, have contact lens Snellen VA equal to or better than 20/30 in each eye.

Exclusion Criteria:

Subjects may not be enrolled in this study if any of the following apply: The subject is/has:

* Wearing lenses in a monovision modality and is unwilling to be fit with distance lenses in both eyes. NOTE: Subjects may not wear lenses in a monovision modality at any time during the study as it will interfere with the visual acuity analysis.
* Poor personal hygiene.
* Any active participation in another clinical trial within 30 days prior to this study.
* Currently pregnant (to the best of the subject's knowledge), is lactating or is planning a pregnancy within the next 3 months.
* A member, relative or household member of the investigator or of the investigational office staff.
* Has a known sensitivity to ingredients used in the over the counter contact lens lubricants approved for use in the study.
* Previous refractive surgery; or current or previous orthokeratology treatment.
* Is aphakic or psuedophakic.
* Ocular or systemic disease such as, but not limited to: anterior uveitis or iritis (past or present), glaucoma, Sjögren's syndrome, lupus erythematosus, sclerodermia, keratoconus or type II diabetes.
* The need for topical ocular medications or any medication which might interfere with contact lens wear or which would require the lenses to be removed during the day.
* The presence of clinically significant (grade 3 or 4) anterior segment abnormalities; inflammations such as iritis; or any infection of the eye, lids, or associated structures.
* A known history of corneal hypoesthesia (reduced corneal sensitivity), corneal ulcer, corneal infiltrates or fungal infections.
* A history of papillary conjunctivitis that has interfered with contact lens wear.
* Slit lamp findings that would contraindicate contact lens wear, including but not limited to:

  * Pathological dry eye or associated dry eye symptoms with decreased tear levels and punctuate staining > Grade 2
  * Pterygium
  * Corneal scars within the visual axis
  * Neovascularization or ghost vessels > 1.0 mm in from the limbus
  * Giant papillary conjunctivitis (GPC) of > Grade 2
  * Anterior uveitis or iritis
  * Seborrheic eczema, seborrheic conjunctivitis or blepharitis

To be eligible to be randomized for study product a subject must have ALL of the Inclusion Criteria and have NONE of the exclusion criteria present.

To be eligible for lens dispensing (either Test or Control), the subject's study lens contact lens visual acuity must be equal to or better than 20/30 in each eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-10; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Byrnes, OD, Principal Investigator; Lee Rigel, OD, Principal Investigator; Mary Jo Stiegemeier, OD, Principal Investigator; Peter Van Hoven, OD, Principal Investigator; Eric White, OD, Principal Investigator
Locations (4):
- United States (4):
  - Eric M. White, OD, Inc., San Diego, California
  - Vision Care Associates, East Lansing, Michigan
  - Western Reserve Vision Care, Beachwood, Ohio
  - Primary Eyecare Group, P.C., Brentwood, Tennessee

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Ninety-three subjects evaluated, 3 subjects found to be ineligible and not randomized or dispensed. 90 adapted single-vision contact lens wearers with myopia were randomized and dispensed on a 2 to 1 ratio within each site and across entire study. Subjects used that same assigned product throughout study duration
Period: Overall Study
Arm/Group | Stenfilcon A Contact Lens | Ocufilcon B Contact Lens
Started | 60 | 30
Completed | 57 | 29
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stenfilcon A Contact Lens | Ocufilcon B Contact Lens | Total
Number analyzed (Participants) | 60 | 30 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 60 | 30 | 90
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.6 (8.884) | 29.8 (8.550) | 31.7 (8.822)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 21 | 59
  Male | 22 | 9 | 31
Region of Enrollment [Number; unit: participants]
  United States | 60 | 30 | 90

OUTCOME MEASURES:

1. Primary Outcome: Objective Assessment: Ocular Response - Biomicroscopy
Description: The primary safety endpoint are the objective slit lamp findings associated with the stenfilcon A contact lenses compared with those same findings reported as associated with the ocufilcon B contact lenses.
  The incidence of biomicroscopy findings (0=not present, 4=severe) over the duration of the study with the highest reported grade was chosen for each unique eye. Biomicroscopy measurements were obtained at Baseline (baseline visit) and All Follow-Ups (week 1 visit, week 2 visit, month 1 visit, month 2 visit combined).The average grade for unique eyes with findings greater than 0 (none) is compared.
Time Frame: Change from baseline visit and all follow-ups visits
Population: Unique eyes are defined as each individual eye in the study and are only counted once for each of the visit groupings
Measure: Mean (Full Range); unit: units on a scale
Units Other Than Participants: unique eyes
Arm/Group | Stenfilcon A Contact Lens | Ocufilcon B Contact Lens
Number analyzed (Participants) | 57 | 29
Number analyzed (unique eyes) | 114 | 58
units on a scale
  Neovascularization, Baseline | 1.00 [1 to 1] | 1.00 [1 to 1]
  Neovascularization, All Follow-up | 1.00 [1 to 1] | 1.10 [1 to 2]
  Corneal Staining, Baseline | 1.00 [1 to 1] | 1.00 [1 to 1]
  Corneal Staining, All Follow-up | 1.09 [1 to 2] | 1.18 [1 to 2]
  Limbal Hyperemia, Baseline | 1.00 [1 to 1] | 1.00 [1 to 1]
  Limbal Hyperemia, All Follow-up | 1.03 [1 to 2] | 1.05 [1 to 2]
  Bulbar Hyperemia, Baseline | 1.00 [1 to 1] | 1.00 [1 to 1]
  Bulbar Hyperemia, All Follow-up | 1.05 [1 to 2] | 1.02 [1 to 2]
  Palperbral Conjunctiva, Baseline | 1.10 [1 to 2] | 1.00 [1 to 1]
  Palpebral Conjunctiva, All Follow-up | 1.38 [1 to 2] | 1.00 [1 to 1]

2. Primary Outcome: Comparison of Objective Findings - Number of Adverse Events in Unique Eyes
Description: The primary safety endpoint in this evaluation will be a comparison of the objective findings of the number of adverse events in unique eyes associated with the stenfilcon A contact lenses compared with those same findings as associated with ocufilcon B contact lenses.
  The number of adverse events over the duration of the study was reported for each unique eye (bilateral or unilateral). Observations for adverse events were reported for any occurrence after dispensing (dispensing visit) through end of month 3 visit (month 3 visit).
Time Frame: Any occurrence from dispensing to month 3 visit
Population: Unique eyes are defined as each individual eye in the study.
Measure: Number; unit: number of adverse events
Units Other Than Participants: unique eyes
Arm/Group | Stenfilcon A Contact Lens | Ocufilcon B Contact Lens
Number analyzed (Participants) | 57 | 29
Number analyzed (unique eyes) | 114 | 58
number of adverse events | 7 | 1

3. Secondary Outcome: Subjective Assessment of Contact Lens Comfort - No Symptoms of Discomfort
Description: The secondary efficacy endpoint is the subjective assessment of contact lens comfort associated with the stenfilcon A contact lens compared with the comfort associated with the ocufilcon B contact lens.
  Subjective comfort assessment is related by the percent number of unique eyes that were reported to have no symptoms of discomfort (0=no symtoms reported) graded on a severity scale of the reported symptoms (0=no symptoms reported, 4=severe) that was experienced over the past month prior to baseline at the baseline visit (Baseline) and any symptoms of discomfort that was experienced since the previous study visit at each scheduled follow-up visit (Week 1, Week 2, Month 1, Month 2, Month 3).
Time Frame: Baseline, Week 1, Week 2, Month 1, Month 2, Month 3
Population: Unique eyes reporting no symptoms of discomfort/Pain, excessive tearing, photophobia, halos, itching/burning, dryness, variable vision, blurred vision, other symptoms.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: unique eyes
Arm/Group | Stenfilcon A Contact Lens | Ocufilcon B Contact Lens
Number analyzed (Participants) | 57 | 29
Number analyzed (unique eyes) | 114 | 58
percentage of eyes
  Baseline | 73.6 | 70.4
  Week 1 | 43.9 | 50.0
  Week 2 | 60.9 | 55.2
  Month 1 | 55.4 | 60.3
  Month 2 | 59.6 | 55.2
  Month 3 | 55.3 | 58.6

4. Primary Outcome: Comparison of Objective Findings for Contact Lens Visual Acuities - Snellen 20/25 VA or Better
Description: The primary efficacy endpoint are the contact lens Snellen visual acuities (VA) of 20/25 VA or better associated with stenfilcon A compared with those same visual acuities associated with ocufilcon B.
  Snellen visual acuity (VA) examinations were performed at All Follow-up visits (week 1 visit, week 2 visit, month 1 visit, month 2 visit). The combined results of All Follow-up visits are compared.
Time Frame: week 1 visit, week 2 visit, month 1 visit, month 2 visit combined
Population: For the completed study subjects, contact lens VA was collected at 562 of the possible 564 examinations (99.6%) for the Test cohort eyes and at 288 of the possible 288 examinations (100%) for the Control cohort eyes.
Measure: Number; unit: percentage of possible examinations
Units Other Than Participants: possible examinations
Arm/Group | Stenfilcon A Contact Lens | Ocufilcon B Contact Lens
Number analyzed (Participants) | 57 | 29
Number analyzed (possible examinations) | 562 | 288
percentage of possible examinations | 99.3 | 100

5. Secondary Outcome: Evaluation of Average Lens Wearing Time - Average Daily Hours Worn
Description: The secondary efficacy endpoint is the objective assessment of the lens average daily wearing times associated with the stenfilcon A compared with the lens average wearing times with the ocufilcon B contact lens. Objective average daily lens wearing time is measured in reported hours worn with the subject's habitual contact lenses recorded at baseline and after dispensing of study lenses recorded at Week 1, Week 2, Month 1, Month 2, Month 3.
Time Frame: Baseline, Week 1, Week 2, Month 1, Month 2, Month 3
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Stenfilcon A Contact Lens | Ocufilcon B Contact Lens
Number analyzed (Participants) | 57 | 29
hours
  Baseline | 15.04 (3.846) | 13.74 (4.182)
  Week 1 | 13.71 (2.281) | 13.18 (2.539)
  Week 2 | 13.69 (2.235) | 13.31 (2.523)
  Month 1 | 13.67 (2.520) | 12.81 (2.640)
  Month 2 | 13.81 (2.774) | 13.41 (2.693)
  Month 3 | 14.00 (2.440) | 13.28 (2.576)

ADVERSE EVENTS:
Arm/Group | Stenfilcon A Contact Lens | Ocufilcon B Contact Lens
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/30
Other Adverse Events (participants affected / at risk) | 3/60 | 0/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stenfilcon A Contact Lens (N=60) | Ocufilcon B Contact Lens (N=30)
Papillary Conjunctivitis (Eye disorders) | 3 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Release of this data (through presentation, publication or other written or oral communication) to other than listed personnel (listed in protocol) requires the prior written permission from the study Sponsor. Study investigators and all office personnel are prohibited from acknowledging participation in the study to individuals and organizations except those listed.